CLINICAL TRIAL: NCT05540470
Title: Radical CUREfor MAlaria Among Highly Mobile and Hard-to-reach Populations in the Guyanese Shield
Acronym: CUREMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Oswaldo Cruz Foundation (Other); Foundation for Scientific Research Suriname (SWOS) Paramaribo, Suriname (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUREMA
Record Dates: First submitted 2022-09-02; First posted 2022-09-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Malaria, Vivax
Keywords: Malaria; Plasmodium vivax; Tafenoquine; Guiana shield; Hard-to-reach populations
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Chloroquine; Primaquine; tafenoquine

STUDY DESIGN:
Intervention Model Description: This is an intervention study, multicentre and international using mixed methods and quasi-experimental design that associates an effectiveness evaluation and an implementation research approach, thus characterising a hybrid design.
  We intend to combine several components that will contribute to achieve the primary and secondary objectives:
  * The intervention per se, which is the core of the study, and combines delivery of the intervention (Module A, Module B or Module A and B) with data collection at inclusion and during a 14-day follow-up.
  * Pre- and post-intervention research (cross-sectional studies), being preponderant for the evaluation of primary objectives (with a quasi-experimental design).
  * A qualitative evaluation of the implementation of the intervention at multiple levels (target population, professionals involved in the study, stakeholders).
  * The modelling study of surveillance data from national malaria programmes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Module A (Experimental): • Module A - PART (Presumptive anti-relapse treatment): This is the core of the strategy for targeting the P. vivax reservoir by identifying individuals with a high probability of being asymptomatic carriers of blood forms and/or hypnozoites (by epidemiological criteria combined with a rapid serological test), and treating these individualswith chloroquine (by 150mgs tablet, according to the following posology: 600mgs on the first day, 450mgs on the second and 300mgs on the third day, or weight-adjusted dosing) and primaquine (in a short regimen of 30 mg per day for seven days, or weight-adjusted dosing) or tafenoquine (300 mg as a single observed dose), after exclusion of contraindications to these treatments. This intervention aims to reduce the likelihood of relapse of a previous infection, and subsequent transmission in forest and urban settings, ultimately helping to reduce the circulation of P. vivax.
  Interventions: Drug: PART
- Module B (Other): • Module B - Malakit: distribution of a self-test and self-treatment kit to individuals in the target population who agree to be trained (and demonstrate understanding of the use of the kit), in order to maintain access to quality test and treatment for malaria attacks that occur in extreme isolation in illegal mining towns in French Guiana
  Interventions: Drug: Malakit
- Pre/post intervention surveys (Other): Two cross-sectional surveys will be conducted in the inclusion sites before and at the end of intervention implementation, during the same period of the year (preferably the last quarter of 2022 and 2024), in order to limit biases associated with seasonality.
  Interventions: Other: CROSS-SECTIONAL PRE- AND POST-INTERVENTION SURVEYS
- QUALITATIVE STUDY (Other): The CUREMA project includes qualitative research that will be conducted before, during and after the intervention by a trained social science researcher. The aim of this research will be to analyse the specific constraints and levers of the intervention under study and the pre-elimination context, in order to draw out lessons that are context-specific but also potentially of universal value. As described above, the study population will be broader and include not only the garimpeiros, but also the study field workers as well as other stakeholders.
  Interventions: Other: QUALITATIVE STUDY

INTERVENTIONS:
Drug: PART — Chloroquine (150mgs tablets) weight-adjusted dosage ; An 8-aminoquinoline drug
  1. Primaquine (PQ) (15 mg tablets): weight-adjusted dosage. Rationale: this short-course posology has been chosen to facilitate the adherence to treatment for asymptomatic individuals participating to the Module A.
     Primaquine will be administered to all participants to Module A during the induction phase of the intervention.
  2. OR tafenoquine (TQ) (150 mg tablets): 2 tablets as a single dose (orally), (Rationale: the posology chosen corresponds to that used in phase III trials for the radical cure of P. vivax and the therapeutic recommendation in Brazil). Tafenoquine will only be administered during the full implementation phase to participants who do not meet exclusion criteria.
  Other Names: chloroquine; primaquine; tafenoquine; module A
  Arms: Module A
Drug: Malakit — delivery of a sturdy, lightweight, waterproof plastic involucre that contains:
  * 1 laminated sheet with illustrated instruction
  * 1 complete anti-malarial treatment targeting P. falciparum, but also effective in acute forms of P. vivax with association with artemisinin derivatives
    * A blister of 24 tablets of Artemether 20 mg + lumefantrine 120 mg of generic medication
    * Two 15 mg tablets of primaquine, to be given as a single dose (145)
  * 1 symptomatic treatment (analgesic, antipyretic): a blister pack of 10 paracetamol 500 mg tablets
  * 3 Malaria rapid diagnostic tests (RDTs) in individual packs and with easy-to-use retractable lancets. Three tests will be included, taking into account the possibility of having one or two negative or invalid tests before returning to a distribution site for further supplies.
  Other Names: module B
  Arms: Module B
Other: CROSS-SECTIONAL PRE- AND POST-INTERVENTION SURVEYS — Surveys will include the collection of a detailed questionnaire on recent malaria and mobility history, a clinical examination, and a venous blood sample
  Other Names: ORPAL 3 - 4
  Arms: Pre/post intervention surveys
Other: QUALITATIVE STUDY — Systematic mapping of stakeholders in the pre-intervention period Semi-structured interviews and focus groups. Observational techniques Participatory approach. Participatory design of a community-based adverse event surveillance system
  Arms: QUALITATIVE STUDY

SUMMARY:
The investigators are proposing a new malaria control strategy to reach the group of garimpeiros not reached by the usual actions of the health services. As it is a complex strategy, several evaluation mechanisms have been designed. The main characteristics of the research are:

* Access to the target population: our target population is represented by miners active and mobile in the south of the Guiana Shield, between Amapá (Brazil), French Guiana (France) and Suriname. To overcome the obstacles posed by the remoteness and clandestinity of the communities of interest, our intervention will take place in the logistical and support hubs (staging areas) of the miners, located in the border regions between the above territories. Thus, it will take advantage of their periodic mobility between these bases and the gold mining sites, and reach the target population where it can be easily accessed.
* The intervention will be combined and will include a common core (malaria health education activity) and two modules that will be offered to participants. Each participant (meeting the inclusion criteria) will be able to choose between participating to one or both modules.

  * The common core of health education will focus on malaria: its causes, means of prevention, the main differences between P. falciparum and P. vivax disease, the importance of a complete treatment against any form of Plasmodium spp.
  * Module A of the intervention will be treatment targeting asymptomatic individuals at risk of carrying P. vivax. The aim of this module is to prevent relapses and reduce the number of human hosts able to transmitthe parasite.
  * Module B of the intervention will correspond to the provision, after appropriate training, of a Malakit self-test and self-treatment kit. The aim of this module is to provide access to quality diagnosis and treatment for episodes of symptoms consistent with malaria that occur in situations of extreme remoteness from health services.
* The purpose of this study is to evaluate a strategy that, if appropriate, can be implemented by health authorities in countries with residual malaria transmission in populations with characteristics similar to our study population. The investigators will therefore use a pragmatic approach so that the conclusions drawn can be transposed as easily as possible to real life, while at the same time putting great effort into the safety of the intervention. Thus, the study field workers who will administer the intervention will have a similar profile to health workers recruited by a large number of malaria control programmes, particularly in remote areas. In addition, monitoring will be simplified and monitoring data can be collected both through face-to-face visits and remotely administered questionnaires.
* The investigators chose to design many of the components of the intervention and study with a participatory approach.
* In order to generate the data necessary for health authorities to potentially take ownership of the intervention in the future, the study will evaluate two aspects of the intervention: effectiveness and implementation.

  * First, the investigators want to evaluate the population-scale effectiveness of the intervention to reduce malaria transmission with a quasi-experimental approach.
  * Secondly, the investigators will analyse the implementation of the intervention, and generate valuable knowledge for further implementation within local health services.

This evaluation will be carried out through the components of the CUREMA study: the intervention itself, pre/post-intervention cross-sectional surveys, the qualitative component and the modelling of epidemiological surveillance data.

• The implementation of these components will have an expected duration of approximately 27 months, the start of inclusions is scheduled for September 2022.

ELIGIBILITY:
Inclusion Criteria for PART and Malakit:

* Be 18 years of age or older
* Agree to participate in the study
* Have an actual involvement in gold mining activities (having been to the garimpo in the last year or planning to enter the garimpo in the following month), regardless of country
* No symptoms of malaria at the time of the inclusion visit
* Weigh over 35 Kg

Eligibility Criteria for PART - Module A -- Wish to take part in module A

- Epidemiological and/or biological criteria in favour of a current asymptomatic carriage of P. vivax (blood stage or liver stage). At least one of the following conditions:

* have a history of clinical malaria during the past 12 months
* OR having a life-long malaria history AND have stayed for at least 1 week during the last 12 months in an area with extensive P. vivax transmission
* OR have a positive P.vivax rapid serological test (if available)

Eligibility Criteria for Malakit - Module B:

* Wish to take part in module B
* Plan to enter agarimpo located in French Guiana the following month

Exclusion Criteria for PART - Module A:

* Refuse to participate in an active follow-up during the 14 days following the start of treatment
* Current pregnancy (declared or rapid urine test positive) or breastfeeding
* Haemoglobinemia below 9 g/dL
* G6PD activity below 70% (for simplicity G6PD activity of 6 UI/dL or below).
* Have received a full course of tafenoquine within the last 3 months or a full course of primaquine in the last month.
* Hypersensitivity or known contraindication to primaquine or tafenoquine or chloroquine
* History of severe mental health disorder
* Being positive for a malaria diagnostic test on the day of inclusion or currently taking anti-malarial treatment.

Exclusion Criteria for Malakit - Module B:

* Inability to self-test (perform and interpret an RDT) during training
* Inability to understand and explain correctly what to do in case of malaria symptoms (tests and ACT posology)

Inclusion criteria for Pre/post intervention surveys

* Be 18 years of age or older
* Agree to participate in the research
* Having left a garimpolocated in French Guiana since maximum one week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1991 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Effectiveness focus | through study completion, an average of 3 years
  To reduce overall the prevalence of symptomatic and asymptomatic infections with Plasmodium spp. as a result of reduced malaria transmission among people involved in gold mining activities in the South of the Guiana Shield
Implementation focus | through study completion, an average of 3 years
  Evaluate the intervention's reach among the target public: reduction in the malaria burden at the collective level in the mining sites and at staging areas

SECONDARY OUTCOMES:
prevalence reduction - Focus on effectiveness | through study completion, an average of 3 years
  To reduce the species-specific prevalence of P. vivax and P. falciparum among people involved in gold mining activities in the South of the Guiana Shield;
contact reduction - Focus on effectiveness | through study completion, an average of 3 years
  To reduce the proportion of garimpeiros with a high probability of recent P. vivax infection (and probably hypnozoite carriers);
malaria incidence reduction - Focus on effectiveness | through study completion, an average of 3 years
  To reduce the incidence of malaria cases associated with gold mining activity in the southern Guyanese Shield, as detected by the epidemiological surveillance systems of the countries involved;
Good use of antimalarial treatment - Focus on effectiveness | through study completion, an average of 3 years
  To increase the proportion of garimpeiros who adequately take anti-malarial treatment when they fall ill in illegal garimpos in French Guiana;
preventing P. vivax parasitaemia - Focus on effectiveness | through study completion, an average of 3 years
  level of P vivax parasietaemia (percentage of red blood cells which contains P. vivax) : estimate the individual-level effectiveness of module A intervention in preventing P. vivax parasitaemia
increase adherence in asymptomatic - Focus on implementation | through study completion, an average of 3 years
  Number of medication taken by the participants related to number of medication delivered to the participants: adherence to the primaquine posology among asymptomatic individuals;
safety - Focus on implementation | through study completion, an average of 3 years
  To assess the safety of medicines for Modules A and B on a community level;
increase health education with specific scales on level of disease comprehension by the participants - Focus on implementation | through study completion, an average of 3 years
  To evaluate the effectiveness of the health education activity carried out during the intervention with specifics scales on level of disease comprehension by the participants;
acceptability of digital tool - Focus on implementation | through study completion, an average of 3 years
  number of participants who regularly use the smartphone application To assess the acceptability of digital tools (smartphone app):
feasability of digital tool - Focus on implementation | through study completion, an average of 3 years
  number of participants who can regularly use the smartphone application:To assess the feasibility of digital tools (smartphone app);
effectiveness of training measured with specifics scales - Focus on implementation | through study completion, an average of 3 years
  Level of comprehension of the training measured with specifics scales: to evaluate the quality and effectiveness of the training received by facilitators;
increase inclusion process - Focus on implementation | through study completion, an average of 3 years
  To assess the fidelity of the inclusion and follow-up process;
quality of rapid serological test - Focus on implementation | through study completion, an average of 3 years
  To evaluate the sensitivity and specificity of the rapid serological test and to estimate the discriminatory capacity of this test to detect recent P. vivax infections in the epidemiological context of the study
intervention's costs measured in euros - Focus on implementation | through study completion, an average of 3 years
  To estimate the programmatic cost of the intervention
needs identification - Focus on implementation | through study completion, an average of 3 years
  highlighting health risk factors by assessing the health situation of garimpeiros and additional health needs beyond malaria elimination
identify facilitating factors and barriers of the intervention - Focus on implementation | through study completion, an average of 3 years
  highlighting the obstacles and levers by assessing facilitating factors as well as barriers to delivering such an intervention in a pre-elimination setting and community involvement to be taken into account for further implementation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Vreden, PhD, Principal Investigator — Foundation for the Advancement of Scientific Research in Suriname; Martha Suaréz-Mutis, PhD, Principal Investigator — Instituto Oswaldo Cruz /IOC /FIOCRUZ
Locations (2):
- Josiane Muller, Oiapoque, Amapá, Brazil
- Stephen vreden, Paramaribo, Suriname, Suriname

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Plessis L, Jimeno Maroto I, Lambert Y, Galindo M, Bardon T, Vreden S, Suarez-Mutis M, Figueira A, Bordalo JM, Douine M, Sanna A. Malaria incubada: a mixed methods analysis on knowledge and experiences on Plasmodium vivax and asymptomatic malaria infections in a hard-to-reach and mobile population in the Amazon. Malar J. 2025 Oct 3;24(1):316. doi: 10.1186/s12936-025-05566-5. PMID 41044665
- [Derived] Douine M, Korsec V, Sanna A, Plessis L, Bardon T, Adenis A, Nacher M, Suarez-Mutis M, Vreden S, Mathieu O, Lambert Y. Prevalence of lead poisoning among artisanal gold miners in French Guiana in 2022: a multicenter cross-sectional observational survey. BMC Public Health. 2025 Aug 14;25(1):2768. doi: 10.1186/s12889-025-24109-w. PMID 40814099
- [Derived] Douine M, Lambert Y, Plessis L, Jimeno I, Galindo M, Bardon T, Le Tourneau FM, Molinie P, Vie A, Adenis A, Nacher M, Figueira da Silva A, Vreden S, Suarez-Mutis MC, Sanna A. Social determinants of health among people working on informal gold mines in French Guiana: a multicentre cross-sectional survey. BMJ Glob Health. 2023 Dec 16;8(12):e012991. doi: 10.1136/bmjgh-2023-012991. PMID 38103896